CLINICAL TRIAL: NCT01702389
Title: Can Opioid-induced Hyperalgesia be Prevented by Gradual Dose Reduction vs. Abrupt Withdrawal of Remifentanil?
Brief Title: Opioid-induced Hyperalgesia After Remifentanil Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marlin Comelon, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011/1639; 2011-002734-39 (EudraCT Number); 11/14666 (Other: Norwegian Medicines Agency)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Hyperalgesia
Keywords: opioid induced hyperalgesia; Pain; Postoperative pain; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia; Pain; Pain, Postoperative | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remifentanil (Experimental): The study has only one arm. Same group of volunteers will receive remifentanil infusion with abrupt withdrawal, remifentanil infusion with gradual dose reduction and saline infusion at three separate trials.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil
  Other Names: Ultiva

SUMMARY:
Remifentanil is a rapid-acting opioid which has been widely used in pain treatment during surgery for the last 15 years 1. Remifentanil is rapidly eliminated (minutes) from the body after end of infusion, and this makes it easily manageable compared to other opioids. However, there are both experimental and clinical studies indicating that remifentanil, after end of infusion, triggers increased pain sensation and increased opioid consumption post-operatively. Increased post-operative opioid consumption should be avoided due to the adverse effects of these drugs (nausea/vomiting, pruritus, dizziness, fatigue and reduced respiratory rate). Thus, it's important to investigate relevant strategies to avoid the increased pain sensation (opioid-induced hyperalgesia = hypersensitivity to pain stimuli) after end of infusion of remifentanil after surgery. Several experimental and clinical trials have been conducted in this field. Ketamine has been shown to block this effect, but its adverse effect profile (i.a. hallucinations) makes it not suitable in normal clinical use. In a study of healthy volunteers, it has been demonstrated that parecoxib (a COX-2 selective NSAID) can prevent remifentanil-induced hyperalgesia. Our group has previously shown that a relatively COX-1 selective NSAID (ketorolac) can prevent hyperalgesia in an experimental pain model.

This is of interest since NSAIDs are frequently administered as premedication before surgery. There are several disadvantages associated with the use of COX-2 inhibitors, e.g. the risk of myocardial infarction after long-term use (> 1 year), and potentially reduced bone healing after orthopedic surgery. However, this has not been shown with short-term use (days/week). The disadvantages associated with the use of e.g. ketorolac (a COX-1 inhibitor) are i.a. increased bleeding tendency, which is unfavourable for the surgeon, and increased risk of gastric ulcer. Therefore, it is of interest to investigate other ways of preventing opioid-induced hyperalgesia. In a recent animal study it has been shown that gradual dose reduction of remifentanil (vs. abrupt withdrawal of a relatively high remifentanil dose) can prevent the development of hyperalgesia after end of infusion. In this study we will i.a. investigate whether this is also the case in humans. In this new model, the study participants will get remifentanil infusion with two different dose reduction regimes: gradual reduction or abrupt withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-60
* Body mass index 17-30
* Healthy volunteers

Exclusion Criteria:

* Use of medication; alternative medicine
* Substance abuse
* Allergies towards medication used in the study
* Participation in other clinical studies the previous 6 months

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hyperalgesia measured by numeric rating scale for pain | 3 weeks
  Two pain models will be used - a heat-pain and a cold-pain model. Testing will be done before, during and after remifentanil infusion. NRS (Numeric rating Scale) will be used for pain scoring.
  Heat model:
  A computer-controlled Medoc ATS Thermal stimulator (3 x 3 cm) is applied to the left volar forearm at pre-defined areas.
  Cold model:
  In the cold test the study participant should keep his right hand in circulating cold water (3 ̊C) in up to 90 seconds.
  The pain models will be applied during three separate trials using remifentanil infusion with abrupt withdrawal, remifentanil infusion with gradual withdrawal and saline infusion(placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Marlin Comelon, MD, Principal Investigator — Oslo UH
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Servin FS. Remifentanil: an update. Curr Opin Anaesthesiol. 2003 Aug;16(4):367-72. doi: 10.1097/01.aco.0000084479.59960.3f. PMID 17021484
- [Background] Angst MS, Koppert W, Pahl I, Clark DJ, Schmelz M. Short-term infusion of the mu-opioid agonist remifentanil in humans causes hyperalgesia during withdrawal. Pain. 2003 Nov;106(1-2):49-57. doi: 10.1016/s0304-3959(03)00276-8. PMID 14581110
- [Background] Hood DD, Curry R, Eisenach JC. Intravenous remifentanil produces withdrawal hyperalgesia in volunteers with capsaicin-induced hyperalgesia. Anesth Analg. 2003 Sep;97(3):810-815. doi: 10.1213/01.ANE.0000078811.80093.88. PMID 12933407
- [Background] Vinik HR, Kissin I. Rapid development of tolerance to analgesia during remifentanil infusion in humans. Anesth Analg. 1998 Jun;86(6):1307-11. doi: 10.1097/00000539-199806000-00033. PMID 9620525
- [Background] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Background] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Background] Koppert W, Sittl R, Scheuber K, Alsheimer M, Schmelz M, Schuttler J. Differential modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by S-ketamine and clonidine in humans. Anesthesiology. 2003 Jul;99(1):152-9. doi: 10.1097/00000542-200307000-00025. PMID 12826855
- [Background] Troster A, Sittl R, Singler B, Schmelz M, Schuttler J, Koppert W. Modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by parecoxib in humans. Anesthesiology. 2006 Nov;105(5):1016-23. doi: 10.1097/00000542-200611000-00024. PMID 17065897
- [Background] Lenz H, Raeder J, Draegni T, Heyerdahl F, Schmelz M, Stubhaug A. Effects of COX inhibition on experimental pain and hyperalgesia during and after remifentanil infusion in humans. Pain. 2011 Jun;152(6):1289-1297. doi: 10.1016/j.pain.2011.02.007. Epub 2011 Mar 10. PMID 21396775
- [Background] Drdla R, Gassner M, Gingl E, Sandkuhler J. Induction of synaptic long-term potentiation after opioid withdrawal. Science. 2009 Jul 10;325(5937):207-10. doi: 10.1126/science.1171759. PMID 19590003
- [Derived] Comelon M, Raeder J, Stubhaug A, Nielsen CS, Draegni T, Lenz H. Gradual withdrawal of remifentanil infusion may prevent opioid-induced hyperalgesia. Br J Anaesth. 2016 Apr;116(4):524-30. doi: 10.1093/bja/aev547. Epub 2016 Mar 1. PMID 26934941